CLINICAL TRIAL: NCT02236975
Title: Prospective, Multi-center, Randomized First-in-man Trial Examining the Safety and Efficacy of BuMA Supreme eG (Electro Grafting) Based Biodegradable Polymer Sirolimus-eluting Stent and Resolute Integrity Zotarolimus-eluting Durable Polymer Stent in Patients With de Novo Coronary Artery Stenosis.
Brief Title: First-in-man Trial Examining the Safety and Efficacy of BuMA Supreme and Resolute Integrity in Patients With de Novo Coronary Artery Stenosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIONEER
Record Dates: First submitted 2014-09-04; First posted 2014-09-11 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2016-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BuMA Supreme Biodegradable drug coating coronary stent system (Experimental): Implant BuMA Supreme stent only
  Interventions: Device: BuMA Supreme Biodegradable drug coating coronary stent system
- Resolute Integrity durable polymer stent system (Active Comparator): Implant Resolute stent
  Interventions: Device: Resolute Integrity durable polymer stent system

INTERVENTIONS:
Device: BuMA Supreme Biodegradable drug coating coronary stent system
  Arms: BuMA Supreme Biodegradable drug coating coronary stent system
Device: Resolute Integrity durable polymer stent system
  Arms: Resolute Integrity durable polymer stent system

SUMMARY:
Prospective, multi-center, randomized 1:1, single blind trial using BuMA Supreme versus Resolute Integrity conducted in approximately 14 interventional cardiology centers in The Netherlands, Belgium, Spain and Portugal.

Clinical follow-up will occur at 1, 9 and 12 months post-stent implantation. All patients will undergo repeat angiography at 9 months follow-up. QCA assessment will be performed at baseline (pre- and post-procedure) and at 9 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is at least 18 years of age.
2. Clinical evidence of ischemic heart disease and/or a positive territorial functional study.
3. Documented stable angina pectoris (Canadian Cardiovascular Society (CCS) Classification 1, 2, 3 or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia
4. The patient has a planned intervention of a single de-novo lesion in one or two separate major epicardial territories (LAD, LCX or RCA).
5. Diameter Stenosis≥50 and<100%.
6. The visually estimated target lesion must be able to be covered by a single BuMA Supreme stent or a single Resolute Integrity stent (for available sizes refer to tables 1 and 2, page 20 and 21).
7. The target lesion reference diameter must be visually estimated to be ≥2.5 mm and ≤4.5 mm in diameter.
8. Written informed consent.
9. The patient agrees to the follow-up visits including a 9 month angiographic follow-up.
10. Patient must have completed the follow-up phase of any previous study.

Exclusion Criteria:

1. Female of child bearing potential (age <50 years and last menstruation within the last 12 months). Subjects with age <50 who underwent tubal ligation, ovariectomy or hysterectomy can be included.
2. Evidence of ongoing acute myocardial infarction (AMI) in ECG and/or elevated cardiac biomarkers (according to local standard hospital practice) have not returned within normal limits at the time of procedure
3. Patient suffered from stroke/TIA during the last 6 months.
4. LVEF <30%
5. Platelet count <100,000 cells/mm3 or >400,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
6. Known renal insufficiency (e.g. serum creatinine >2.5mg/dL, or creatinine clearance ≤30 mL/min), or subject on dialysis, or acute kidney failure (as per physician judgment).
7. Patient undergoing planned surgery within 6 months with the necessity to stop DAPT.
8. Patient requiring oral anticoagulation (Coumadin, Novel Oral Anticoagulant (NOAC))
9. History of bleeding diathesis or coagulopathy
10. The patient is a recipient of a heart transplant
11. Known hypersensitivity or contraindication to aspirin, heparin, antiplatelet medication specified for use in the study, sirolimus, zotarolimus, or cobalt-chromium.
12. Other medical illness (e.g. cancer, stroke with neurological deficiency) or known history of substance abuse (alcohol, cocaine, heroin etc.) as per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy
13. The patient is simultaneously participating in another investigational device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss | Up to 9 month
  The primary endpoint is in-stent Late Lumen Loss (LLL) at 9 months after stent implantation as assessed by off-line QCA.

SECONDARY OUTCOMES:
Angiographic endpoint | 9 and 12 month
  Acute Lumen Gain (mm);
Angiographic endpoint | 9 and 12 month
  MLD (mm) post procedure and at 9 months;
Angiographic endpoint | 9 and 12 month
  Diameter Stenosis (%) post procedure and at 9 months;
Angiographic endpoint | 9 and 12 month
  Binary Restenosis (DS ≥50%) at 9 months
Clinical endpoint | 9 and 12 month
  Acute success (device and procedural success)
Cinical endpoint | 9 and 12 month
  Device-oriented Composite Endpoints (DoCE) at 1, 9 and 12 months and its individual components. (Device-oriented Composite Endpoint is defined as Cardiac Death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated Target Lesion Revascularization).
Clinical endpoint | 9 and 12 month
  Myocardial infarction (Q-wave, Non q-wave) at all time points.
Clinical endpoint | 9 and 12 month
  Any revascularization at all time points.
Clinical endpoint | 9 and 12 month
  Stent thrombosis according to the ARC definitions up to 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens von.Birgelen, MD,Phd, Principal Investigator — Medisch Spectrum Twente (MST), Enschede, the Netherlands; Manel Sabate, MD,Phd, Principal Investigator — Clinic university hospital Barcelona, Spain; Patrick W.Serruys, MD,Phd, Study Chair — Interventional Cardiology, Thorax center, Erasmus MC, Rotterdam
Locations (12):
- Belgium (3):
  - Imelda Hospital, Bonheiden
  - CHU Chaleroi, Chaleroi
  - Oost-limburg Hospital, Genk
- Netherlands (4):
  - AMC, Amsterdam
  - OLVG, Amsterdam
  - UMCG, Groningen
  - Maasstad Hospital, Rotterdam
- Portugal (3):
  - Hospita; Garcia de Orta, Almada
  - Santa Maria University Hospital, Lisbon
  - Gaia/Espinho Hospital Centers, Porto
- Spain (2):
  - University Hospital Madrid, Madrid
  - Hospital Álvaro Cunqueiro, Vigo

REFERENCES:
- [Derived] Wang R, Kawashima H, Hara H, Gao C, Ono M, Takahashi K, Tu S, Soliman O, Garg S, van Geuns RJ, Tao L, Wijns W, Onuma Y, Serruys PW. Comparison of Clinically Adjudicated Versus Flow-Based Adjudication of Revascularization Events in Randomized Controlled Trials. Circ Cardiovasc Qual Outcomes. 2021 Nov;14(11):e008055. doi: 10.1161/CIRCOUTCOMES.121.008055. Epub 2021 Oct 20. PMID 34666500